CLINICAL TRIAL: NCT02428907
Title: Simulation Based Team Training of Endoscopy Staff May Improve Patients' Perception of Colonoscopy
Brief Title: Simulation Training of Endoscopy Staff to Improve Patient Experience in Colonoscopy
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-58-0028
Record Dates: First submitted 2015-02-18; First posted 2015-04-29 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
Keywords: simulation training; minimal sedation; colonoscopy; patient satisfaction; teamwork; team training; patient safety
MeSH Terms: conditions — Colorectal Neoplasms; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: simulation training — teamtraining of endoscopy staff

SUMMARY:
Some patients experience a degree of pain and discomfort during endoscopic examination of the large bowel. Sedatives and analgesics may be administered in low doses. Excessive dosage or intense pain may lead to hypotension and impaired level of consciousness. The purpose of the present study was to determine if simulation training of endoscopy staff in preventing pain and handling acute complications through effective teamwork could improve the quality of colonoscopy from the patients' perspective.

DETAILED DESCRIPTION:
The study was carried out in a surgical department, where colonoscopies were performed on an out-patient basis under minimal sedation. The intervention consisted of a simulation based course for endoscopy staff. All endoscopy nurses and doctors participated (n=43). The course consisted of three short lectures followed by simulation training. The lectures dealt with technical aspects of colonoscopy, usage of medication and management of unexpected emergency events during the procedure, and finally with interprofessional teamwork and team communication. The lectures were followed by in situ simulation in an endoscopy room. For 2 months before and after the course a questionnaire based survey was carried out. The respondents were consecutive patients who had undergone colonoscopy under minimal sedation or no sedation (according to their own preference ). The questionnaire was filled out when the patient was fully recovered after sedation and ready to go home. The relevant nursing staff and doctor for the procedure also filled out their part of the questionnaire. Patients were invited to participate and gave written consent after oral and written information according to the Helsinki declaration .

ELIGIBILITY:
Inclusion Criteria:

* All patients for colonoscopy under minimal sedation who are able to understand imformation

Exclusion Criteria:

* Unable to understand information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for colonoscopy under minimal sedation
Sampling Method: Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
patient perception of colonoscopy | 3 months
  comparison of patient satisfaction aspects of colonoscopy before and after a simulation, course for staff. The patients fill out a questionnaire: Pain score on a visual analogue scale, Wiilingness to return for a repeat colonoscopy if necessary on a visual analogue scale, assessmment of doctor's and nurse's behaviour on a scale from 1 - 10 regarding empathy, quality of information. Staff answer a questionnaire where they assess the quality of teamwork on a scale from 1-10. They also assess the patients perceived pain on a visual analogue scale.

SECONDARY OUTCOMES:
Staff perception of teamwork | 3 months
  comparison of staff's perception of quality of teamwork before and after a simulation course

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Larsen, m.d., Principal Investigator — Medical Doctor and head of department at Aalborg University Hospital
Locations (1):
- NordSim, Aalborg University Hospital, Aalborg, Denmark